CLINICAL TRIAL: NCT05439447
Title: A Study on Building a Voice Cohort for the Development of a Non-face-to-face Machine Learning Diagnostic and Monitoring Platform Using Voice Analysis and Various Sensors in Patients With Dysphagia.
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Other Study IDs: B-2206-761-302
Record Dates: First submitted 2022-06-16; First posted 2022-06-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for VFSS examination due to dysphagia.
  Interventions: Diagnostic Test: Patients scheduled for VFSS testing group

INTERVENTIONS:
Diagnostic Test: Patients scheduled for VFSS testing group — Patients scheduled for VFSS testing, patient with voice.

SUMMARY:
Collection of basic data for real-time analysis and monitoring by measuring what changes in voice occur according to the state of dysphagia using voice analysis and various sensors.

DETAILED DESCRIPTION:
* Design : Prospective cohort study
* Setting : Hospital rehabilitation department
* Inclusion criteria of the patient group : Patients scheduled for VFSS examination
* Intervention

  * This study will be conducted after collecting basic information such as age, gender, and disease of patients who met the inclusion criteria among patients scheduled to undergo a video fluoroscopic swallowing test (VFSS test) for the diagnosis of dysphagia, and after obtaining guidance and consent through the study description will do.
  * Before the subject's VFSS test, "Ah for 5 seconds", after clearing the throat, "Ah for 5 seconds", and briefly cut with a slightly high sound, "Ah. oh Ah.", shut lips lightly and read "Ummm~~~~", read a short sentence.
  * While the subject makes the above sound, voice is recorded, video is taken, and integrated sensors such as a microphone (sound detection) sensor and surface electromyography sensor are attached to measure changes in each sensor.
  * After the VFSS test, participants will repeat the above sound and record the same twice. (As before the test, imaging of the patient's swallowing is also performed.)
  * Using voice analysis, various sensor values, and image information, a voice indicator that can predict the amount of suction and residue on the VFSS test is found.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years of age or older and do not fall under the exclusion criteria
* Patients scheduled for VFSS test
* Patients who can record voices such as "Ah.", "Ummm~~~", short sentences
* Patients who can attach sensor on their throat
* Those who voluntarily consent to the clinical trial

Exclusion Criteria:

* Those who do not agree to participate in this study
* Patients who can not follow Step 1 instructions
* Patients who can not vocalize or follow to speak
* Patients who cannot apply the sensor due to skin allergy or hypersensitivity to sensor attachment
* Other who have comorbidities (e.g., maligant tumors, blood clotting abnormalities, etc.) that are inappropriate for clinical trial participation by the judgment of the researcher 6) Other who are judged by the researcher to be unsuitable for this clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for VFSS examination due to dysphagia
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Voice analysis before and after meals, the results are compared with VFSS to verify significant indicators (residue, aspiration, etc.) by Paired t-test analysis. | Baseline/ Change from baseline when swallowing
  By comparing the VFSS swallow test result with the analysis value through voice analysis, the accuracy of the case classified as aspiration in the voice test is used as the primary indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, M.D, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No